CLINICAL TRIAL: NCT04165018
Title: Prospective Study FNB, Is It Time To Abandon Cytological Assessment (FACET)
Brief Title: Prospective Study FNB, Is It Time To Abandon Cytological Assessment
Acronym: (FACET)
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-44963
Record Dates: First submitted 2019-11-01; First posted 2019-11-15 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic masses and lesions
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Biospecimen Retention: Samples Without DNA — Pancreatic mass biopsy for pathological evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Fine-Needle Biopsy (FNB) — Fine-needle biopsy may be used to take samples of a pancreatic neoplasm.

SUMMARY:
Endoscopic Ultrasound (EUS) is a minimally invasive procedure used by gastroenterologists to examine pancreatic masses and lesions. A fine needle is traversed through an endoscope and used to acquire tissue samples, which are then sent for pathology. The standard approach for diagnosing solid pancreatic lesions has been fine needle aspiration (FNA) (Han et al. 2016). However, the use of FNA comes with its limitations, some of which include multiple needle passes to acquire fluid, the need for on-site cytologists, and decreased diagnostic yield. Fine needle biopsy (FNB) is the latest approach being employed by endosonographers in lieu of FNA. FNB confers several advantages over FNB. First, FNB requires fewer needle passes than FNA to acquire tissue sample for immunohistochemical staining. In addition, FNB provides better tissues samples, greater sensitivity of the tissue core, and thus, improved diagnostic yields (Tian et al. 2018). Finally, FNB is more cost-effective than FNA and relies on pathologists, instead of on-site cytologists, and preserves the tissue core (Tian et al. 2018). The objective of this study is to establish a database of samples placed in formalin for patients who will undergo a fine-needle biopsy (FNB) for pathological evaluation without rapid on site cytological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than or equal to 18 years of age
* Patient is referred to EUS-FNB for pancreatic mass lesions

Exclusion Criteria:

* Patient is younger than 18 years of age
* Patient refused and/or unable to provide consent
* Patient is a pregnant woman

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred to EUS-FNB for pancreatic mass lesions
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity using FNB sampling pancreatic mass | 2 years
  % of core tissue obtained, number of needle passes made, and assessment of any procedure related adverse events
Diagnostic yield between FNB samples placed in formalin for pathology evaluation from two different types of needle | 2 years

SECONDARY OUTCOMES:
Rate of adverse events of utilizing the FNB technique, including pancreatitis, bleeding, or perforation | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Lukes Medical Center (BSLMC), Houston, Texas